CLINICAL TRIAL: NCT00066326
Title: Phase I Study Of The Combination Of 17-AAG And Imatinib Mesylate (Gleevec) In Patients With Blastic Phase, Accelerated Phase Of Chronic Mesylate Leukemia (CML) Or Patients With Chronic Phase CML Who Have Not Achieved A Cytogenetic Response With Imatinib Mesylate
Brief Title: Imatinib Mesylate and 17-N-Allylamino-17-Demethoxygeldanamycin in Treating Patients With Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000315521; U01CA062487 (NIH); P30CA022453 (NIH); WSU-C-2599; NCI-5932
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Leukemia
Keywords: blastic phase chronic myelogenous leukemia; Philadelphia chromosome positive chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase | interventions — Imatinib Mesylate; tanespimycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: imatinib mesylate
Drug: tanespimycin

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth. Drugs used in chemotherapy such as 17-N-allylamino-17-demethoxygeldanamycin use different ways to stop cancer cells from dividing so they stop growing or die. Combining imatinib mesylate with chemotherapy may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of 17-N-allylamino-17-demethoxygeldanamycin when given together with imatinib mesylate in treating patients with chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose-limiting toxicity of 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) when administered with imatinib mesylate in patients with chronic myelogenous leukemia.
* Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is an open-label, nonrandomized, multicenter, dose-escalation study of 17-N-allylamino-17-demethoxygeldanamycin (17-AAG).

Patients receive oral imatinib mesylate on days 1-21 and 17-AAG IV over 1 hour on days 1, 4, 8, and 12. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of 17-AAG until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional cohort of 6-10 patients receives treatment at the recommended phase II dose.

PROJECTED ACCRUAL: Approximately 21-42 patients will be accrued for this study within 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic myelogenous leukemia, including any of the following phases:

  * Blastic phase

    * Greater than 30% blasts in the peripheral blood or bone marrow
    * Previously untreated disease OR refractory to or relapsed after most recent therapy
  * Accelerated phase, defined by 1 of the following:

    * At least 15, but less than 30%, blasts in the peripheral blood or bone marrow
    * At least 30% blasts and promyelocytes in the peripheral blood or bone marrow
    * Greater than 20% peripheral blood basophilia
  * Chronic phase

    * No major cytogenetic response (less than 65% Philadelphia chromosome negative) after 12 months of prior imatinib mesylate therapy
* Philadelphia chromosome positive by routine cytogenetics

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* ALT and AST no greater than 2.5 times upper limit of normal

Renal

* Creatinine less than 1.5 mg/dL

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known allergy to eggs
* Able to swallow pills
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent uncontrolled medical illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior stem cell transplantation

Chemotherapy

* More than 4 weeks since prior chemotherapy (except hydroxyurea or anagrelide) (at least 6 weeks for nitrosoureas or mitomycin)

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy

Surgery

* No prior liver, kidney, or lung transplantation
* More than 14 days since prior major surgery (e.g., thoracotomy or intra-abdominal surgery)

Other

* Prior imatinib mesylate administered within the past 4 weeks is allowed
* No concurrent tacrolimus or cyclosporine as immunosuppressive agents
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent agents that alter CYP3A4 activity, including any of the following:

  * Grapefruit juice
  * Ketoconazole
  * Fluconazole
  * Itraconazole
  * Erythromycin
  * Clarithromycin
  * Cimetidine
  * Terfenadine
  * Astemizole
  * HIV protease inhibitors (e.g., indinavir and nelfinavir)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-06; Primary Completion 2004-10 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles A. Schiffer, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States